CLINICAL TRIAL: NCT02280694
Title: Metronomic Poly-chemotherapy for Metastatic Colorectal Cancer at Progression Following Established Treatments: Clinical and Laboratory Research
Brief Title: Low Dose Metronomic Poly-chemotherapy for Metastatic CRC
Acronym: LDMchemoCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0035-14-EMC
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Cyclophosphamide; Methotrexate; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- capecitabine, cyclophosphamide, methotrexate, celecoxib (Experimental): The Investigational Product: Route and Dosage Form Ambulatory/oral, continuous but not uniform, DAILY treatment
  1. Tab. CYCLOPHOSPHAMIDE 50mg, 1X1/day ONLY days 1-5 / week; At evening only (at the end of meal)
  2. Tab. CAPECITABINE 500mg, fixed dose of 1500mg/day (1000mg at morning + 500mg at evening) ONLY on days 1-5 / week; At morning AND at evening (at the end of meals)
  3. Tab. METHOTREXATE 2.5mg, 1x2/day ONLY on days 6-7/week; At morning AND evening (one hour before meal)
  4. Tab. CELECOXIB 200 mg, 1x2/day EVERY day (at the end of meal)
  Interventions: Drug: Capecitabine; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Celecoxib

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
Drug: Cyclophosphamide
  Other Names: Endoxan
Drug: Methotrexate
  Other Names: Abitrexate, Methotrexat "Ebewe", Metoject medac
Drug: Celecoxib
  Other Names: Celebra, Celcox

SUMMARY:
This study investigates the activity of a new regimen of treatment for patients with metastatic colorectal carcinoma. This includes a combination of well-known chemotherapy agents and anti-inflammatory agents, when administered orally at low daily doses and without planed brakes (Low Dose Metronomic regimen), in contrast with the conventional and already exhausted regimens of treatment at Maximal Tolerated Doses (MTD) which required pre-planned brakes between treatment days.

DETAILED DESCRIPTION:
Patients suffering from metastases of colorectal cancer whose tumor cells develop resistance to conventionally administered treatments are in need for new methods of treatment.

While their chemotherapy had been administered up till then at the classical regimen of Maximal Tolerated Doses (MTD), which is aimed to directly killing maximal fractions of tumor cells, the present study evaluates the clinical benefit of a treatment which is based on old chemotherapeutic and old anti-inflammatory drugs, when these are administered at low doses,on daily basis and orally taken, without planed brakes (Low Dose Metronomic regimen).

Treatments based on this type of regimen have already been studied on other models of cancer and showed the capacity of suppressing tumor growth by a new category of anti-tumor effects. Namely, by affecting factors and mechanisms which prevail in the microenvironment that surrounds tumor deposits, thus circumventing the resistance of their cancer cells to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological (or cytological) proof of colorectal carcinoma (CRC)
2. Measurable metastases
3. ECOG (Eastern Cooperative Oncology Group) performance status 0-2
4. Progressing disease following all available chemotherapy treatment lines (including chemotherapy, bevacizumab+/-ziv-aflibercept, and an epidermal growth factor receptor (EGFR) inhibitor [if WT(wild type)-KRAS]
5. The central-radiologist's confirmation of PD* under the last (previous) line of "conventional treatment".

   * PD (progressive disease) by RECIST(Response Evaluation Criteria in Solid Tumors) criteria : a) there is 20% or more relative increment in the sum of diameters of target lesions in comparison with the base line sum, and their absolute increase is 5 mm. or more, or b) there appeared one or more new lesions, or c)there is substantial worsening in non-target disease
6. Age: between 18 and 85
7. Prior radiotherapy either as adjuvant treatment or for palliation is allowed, unless this was delivered to the only measurable lesion
8. Complete blood count reflecting adequate Bone Marrow:

Hb=/ > 9 g/dL, ANC=/> 1,500 Plt =/> 75,000/mcL; 9. Adequate liver function:

1. Total Bilirubin always =/<X1.5 ULN
2. ALT and AST and Alkaline Phosphatase =/ < 2.5 X upper normal limit , although in patients with liver metastases these are acceptable if =/< 5 X ULN; 11. Adequate renal function (serum creatinine): =/< 1.5 X ULN. 12. Absence of any non-hematological toxicity at grade 2 or higher. 13.The patient is able to understand and ready to sign the informed consent

Exclusion Criteria:

1. Lack of confirmation of PD (under the pre-study treatment) by the central radiologist
2. Any concurrent other active cancer (except basal cell or squamous cell carcinoma of skin and early prostate cancer or DCIS- in situ breast cancer)
3. Inability to adhere to monthly visits to the oncological unit for evaluation
4. Presence of brain metastases
5. Continuous treatment with steroids or with NSAIDs or with anticoagulants during the last year (except micropirin)
6. Previous radiotherapy to the only site of measurable disease
7. Existence of active peptic ulcer or symptomatic coronary disease
8. Existence of chronic inflammatory diseases, such as ulcerative colitis or Crohn's disease or rheumatoid arthritis
9. Presence of ascites, and/or any other "third space" finding (eg. significant leg edema)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The median progression free survival (mPFS) | Base line and every consecutive 8 weeks, up to disease progression or exit from study for any other cause, up to 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Purim, MD, Principal Investigator — Gastrointestinal Oncology Unit, Institute of Oncology, Davidoff Center, Rabin Medical Center, Belinson Campus, Petach Tiqva, Israel
Locations (1):
- Gastrointestinal Oncology Unit, Institute of Oncology, Davidoff Center, Rabin Medical Center, Belinson Campus,, Petach Tiqva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Von Hoff DD, Stephenson JJ Jr, Rosen P, Loesch DM, Borad MJ, Anthony S, Jameson G, Brown S, Cantafio N, Richards DA, Fitch TR, Wasserman E, Fernandez C, Green S, Sutherland W, Bittner M, Alarcon A, Mallery D, Penny R. Pilot study using molecular profiling of patients' tumors to find potential targets and select treatments for their refractory cancers. J Clin Oncol. 2010 Nov 20;28(33):4877-83. doi: 10.1200/JCO.2009.26.5983. Epub 2010 Oct 4. PMID 20921468